CLINICAL TRIAL: NCT00423488
Title: A Multicenter, Randomized, Parallel-Groups, Double-Blind Placebo Controlled Study Comparing the Efficacy, Safety, and Tolerability of Co-administration of Ezetimibe 10 mg With Ongoing Treatment With Simvastatin 20 mg Versus Doubling the Dose of Simvastatin in Subjects With Primary Hypercholesterolemia Diabetes Mellitus Type 2 and Coronary Heart Disease
Brief Title: Ezetimibe and Simvastatin in Primary Hypercholesterolemia, Diabetes Mellitus Type 2, and Coronary Heart Disease (COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04037
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Diabetes Mellitus, Type 2; Coronary Disease
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus, Type 2; Coronary Disease | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg (Experimental): Participants were instructed to take one 10-mg ezetimibe tablet and one simvastatin placebo tablet orally in the evening every day for six weeks in addition to their daily, oral, open-label, 20-mg simvastatin tablet.
  Interventions: Drug: Ezetimibe 10 mg; Drug: Simvastatin 20 mg; Drug: Simvastatin Placebo
- Ezetimibe Placebo + Simvastatin 40 mg (Active Comparator): Participants were instructed to take one ezetimibe placebo tablet and one simvastatin 20-mg tablet orally in the evening every day for six weeks in addition to their daily, oral, open-label, 20-mg simvastatin tablet.
  Interventions: Drug: Simvastatin 20 mg; Drug: Ezetimibe Placebo

INTERVENTIONS:
Drug: Ezetimibe 10 mg — 1 x 10-mg tablet, provided as blinded study treatment
  Arms: Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg
Drug: Simvastatin 20 mg — 1 x 20-mg tablet, provided as open-label study treatment
Drug: Ezetimibe Placebo — 1 tablet matching ezetimibe 10-mg tablet, provided as blinded study treatment
  Arms: Ezetimibe Placebo + Simvastatin 40 mg
Drug: Simvastatin 20 mg — 1 x 20-mg tablet, provided as blinded study treatment
  Arms: Ezetimibe Placebo + Simvastatin 40 mg
Drug: Simvastatin Placebo — 1 tablet matching 20-mg simvastatin tablet, provided as blinded study treatment
  Arms: Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will assess, after 6 weeks of dosing, whether co-administration of ezetimibe 10 mg with simvastatin 20 mg will be more effective than treatment with doubling the dose of simvastatin to 40 mg alone in reducing low-density lipoprotein-cholesterol (LDL-C) concentrations and in achieving the National Cholesterol Expert Panel (NCEP) III LDL-C target goal of <2.6 mmol/L (<100 mg/dL) for subjects with diabetes mellitus and coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have diabetes mellitus type 2 (fasting plasma glucose >7 mmol/L [126 mg/dL]) of at least 12 months duration at Visit 3 and must be adequately controlled (glycated hemoglobin [HbA1c] <=9.0%). Subjects must not have had a change in antidiabetic pharmacotherapy [i.e. changes in dosage (with the exception of +/- 10 units of insulin) or addition of new medication] or experience recent history of repeated hypoglycemia or unstable glycemic control within 3 months of Visit (Baseline Visit).
* Subjects must have documented coronary heart disease (CHD). For the purposes of this study, CHD will include one or more of the following features: documented stable angina with evidence of ischemia on exercise testing); history of myocardial infarction; history of percutaneous transluminal coronary intervention (PCTI) with or without stent placement); symptomatic peripheral vascular disease (claudication); documented history of atherothrombotic cerebrovascular disease; and/or documented history of unstable angina or non-Q wave myocardial infarction.
* Subjects must have a low-density lipoprotein cholesterol (LDL-C) concentration >=2.6 mmol/L (100 mg/dL) to <=4.1 mmol/L (160 mg/dL) using the Friedewald calculation available at the time of randomization Visit 3 (Baseline Visit).
* Subjects must have triglyceride concentrations of <3.99 mmol/L (350 mg/dL) at Visit 3 (Baseline Visit).
* Subject must be currently taking simvastatin 20 mg daily and by history has taken 80% of daily evening doses for the 6 weeks prior to Visit 3 (Baseline Visit).
* Subject must be >=18 years and <=75 years of age.
* Subjects must have maintained a cholesterol lowering diet and exercise program for at least 4 weeks prior to Screening (Visit 2) and be willing to continue the same diet and exercise program during the study.
* Subjects must have liver transaminases (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) <50% above the upper limit of normal, with no active liver disease, and creatinine kinase (CK)<50% above the upper limit of normal at Visit 3 (Baseline Visit).
* Clinical laboratory tests (complete blood count (CBC), blood chemistries, urinalysis) must be within normal limits or clinically acceptable to the investigator at Visit 3 (Baseline Visit).
* Subjects must report a stable weight history for at least 4 weeks prior to entry into study at Visit 3 (Baseline Visit).
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, must have been maintained on a stable dose and regimen for at least 8 weeks and be willing to continue the same regimen for the duration of the study.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically-prescribed intrauterine device (IUD), condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must be free of any clinically significant diseases other than diabetes mellitus or coronary heart disease that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and must agree to remain on their cholesterol-lowering diet and their exercise regimen for the duration of the study
* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.

Exclusion Criteria:

* Subjects whose body mass index (BMI = weight[kg]/height[m]**2) is >=35 kg/m**2 at Visit 3 (Baseline Visit).
* Subjects who consume >14 alcoholic drinks per week. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Any condition or situation which, in the opinion of the investigator, might pose a risk to the subject or interfere with participation in the study.
* Women who are pregnant or nursing.
* Congestive heart failure defined by New York Heart Association (NYHA) as Class III or IV.
* Uncontrolled cardiac arrhythmia.
* Myocardial infarction, acute coronary insufficiency, coronary artery bypass surgery, or angioplasty within 3 months of Visit 3 (Baseline Visit).
* Unstable or severe peripheral artery disease within 3 months of Visit 3 (Baseline Visit).
* Newly diagnosed or currently unstable angina pectoris.
* Uncontrolled hypertension (treated or untreated) with systolic blood pressure >160 mmHg or diastolic >100 mmHg at Visit 3 (Baseline Visit).
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, i.e., secondary causes of hyperlipidemia, such as secondary hypercholesterolemia due to hypothyroidism (thyroid stimulating hormone [TSH] above upper limit of normal) at Visit 3. Subjects with a history of hypothyroidism who are on a stable therapy of thyroid hormone replacement for at least 6 weeks are eligible for enrollment if TSH levels are within normal limits at Visit 3 (Baseline Visit).
* Impaired renal function (creatinine >2.0 mg/dL) or nephrotic syndrome at Visit 3 (Baseline Visit).
* Disorders of the hematologic, digestive, or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Known human immunodeficiency virus (HIV) positive.
* Cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Subjects who have not observed the designated wash-out period for any of the prohibited medications.
* Subjects currently consuming large amounts of grapefruit juice (>1 liter/day).
* Oral corticosteroids, unless used as replacement therapy for pituitary/adrenal disease and the subject is on a stable regimen for at lest 6 weeks prior to Visit 3 (Baseline Visit).
* Subjects who are currently using cardiovascular medication (e.g., antihypertensive, antiarrhythmic) and have not been on a stable regimen for at least 6 weeks prior to Visit 3 (Baseline Visit) and it is expected to change during the study.
* Subjects who are currently using psyllium, other fiber-based laxatives, and/or any other over-the-counter (OTC) therapy known to affect serum lipid levels (phytosterol margarine), and have not been on a stable regimen for at least 5 weeks prior to study entry Visit 3 (Baseline Visit) and who do not agree to remain on this regimen throughout the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-07-12 (Actual); Primary Completion 2007-02-16 (Actual); Study Completion 2007-02-16 (Actual)

REFERENCES:
- [Result] Bardini G, Giorda CB, Pontiroli AE, Le Grazie C, Rotella CM. Ezetimibe + simvastatin versus doubling the dose of simvastatin in high cardiovascular risk diabetics: a multicenter, randomized trial (the LEAD study). Cardiovasc Diabetol. 2010 May 21;9:20. doi: 10.1186/1475-2840-9-20. PMID 20492655
- [Derived] Rotella CM, Zaninelli A, Le Grazie C, Hanson ME, Gensini GF. Ezetimibe/simvastatin vs simvastatin in coronary heart disease patients with or without diabetes. Lipids Health Dis. 2010 Jul 27;9:80. doi: 10.1186/1476-511X-9-80. PMID 20663203

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg: Participants were instructed to take one 10-mg ezetimibe tablet and one simvastatin placebo tablet orally in the evening every day for six weeks in addition to their daily, oral, 20-mg simvastatin tablet.
- Ezetimibe Placebo + Simvastatin 40 mg: Participants were instructed to take one ezetimibe placebo tablet and one simvastatin 20-mg tablet orally in the evening every day for six weeks in addition to their daily, oral, 20-mg simvastatin tablet.
Period: Overall Study
Arm/Group | Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg | Ezetimibe Placebo + Simvastatin 40 mg
Started | 42 | 51
Completed | 37 | 50
Not Completed | 5 | 1
Not completed — No evidence of study drug intake | 2 | 1
Not completed — No post baseline data | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg | Ezetimibe Placebo + Simvastatin 40 mg | Total
Number analyzed (Participants) | 42 | 51 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (6.5) | 63.9 (6.1) | 64.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 24 | 39 | 63
Region of Enrollment [Number; unit: participants]
  Italy | 42 | 51 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Endpoint, After 6 Weeks of Treatment
Time Frame: 6 weeks of treatment (from Baseline to Endpoint)
Population: Intent-to-treat population only.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg | Ezetimibe Placebo + Simvastatin 40 mg
Number analyzed (Participants) | 37 | 50
percentage change | -32.2 (15.7) | -20.8 (20.1)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg vs Ezetimibe Placebo + Simvastatin 40 mg; Test type: Superiority or Other; p = 0.005, ANOVA; The analysis of variance (ANOVA) model included term of treatment effect. If more than one basal value was available, the latest was used; least-squares means = -11.5, 95% CI [-19.4 to -3.5]

ADVERSE EVENTS:
Description: The ezetimibe 10 mg + simvastatin placebo + simvastatin 20 mg safety population is comprised of 40 subjects as there was no evidence of study drug intake for 2 of the 42 randomized. The ezetimibe placebo + simvastatin 40 mg safety population is comprised of 50 participants as there was no evidence of study drug intake for 1 of the 51 randomized.
Arm/Group | Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg | Ezetimibe Placebo + Simvastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/50
Other Adverse Events (participants affected / at risk) | 0/40 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe 10 mg + Simvastatin Placebo + Simvastatin 20 mg (N=40) | Ezetimibe Placebo + Simvastatin 40 mg (N=50)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish or publicaly present results without prior written authorization from the sponsor, except than for the dispositions provided for in Ministerial Circular n.6 of 02 SEP 2002 and, particularly, disposition n.1a) The investigator further agrees to provide 30 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of material(including text for oral presentation) that report study results.